CLINICAL TRIAL: NCT00465894
Title: Randomized Controlled Trial of Tolterodine in Combination With or Without Low-Dose Intravaginal Estradiol Cream for the Treatment of Overactive Bladder in Post-Menopausal Women
Brief Title: Detrol Long Acting (LA) vs Estrace Vaginal Cream for the Treatment of Overactive Bladder Symptoms
Acronym: DRIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, David Rich Ellington, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F061208008; IIR - DRIVE
Record Dates: First submitted 2007-04-23; First posted 2007-04-25 (Estimated); Results first posted 2012-10-23 (Estimated); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Overactive Bladder
Keywords: overactive bladder; urge leakage; nightime urination; incontinence; urinary frequency
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Tolterodine Tartrate; Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Extended Release Tolterodine LA (Active Comparator): An anti-muscarinic drug that is used for symptomatic treatment of urinary incontinence.
  Interventions: Drug: Extended Release Tolterodine LA
- Intra Vaginal Estradiol Cream (Active Comparator): For topical application to the vaginal area to treat symptoms of urgency or irritation with urination.
  Interventions: Drug: Intra Vaginal Estradiol Cream

INTERVENTIONS:
Drug: Extended Release Tolterodine LA — Tolterodine LA 4 mg once daily for 52 weeks. At 12 Weeks, the subjects were offered the addition of the alternative therapy with follow-up at 24 and 52 weeks
  Other Names: Detrol
  Arms: Extended Release Tolterodine LA
Drug: Intra Vaginal Estradiol Cream — 17-B estradiol cream 0.5 grams nightly for 6 weeks then two times weekly for 46 weeks. At 12 Weeks, the subjects were offered the addition of the alternative therapy with follow-up at 24 and 52 weeks.
  Other Names: Estrace; Premarin vaginal cream
  Arms: Intra Vaginal Estradiol Cream

SUMMARY:
The purpose of this study is to determine if long acting tolterodine confers more benefit than intravaginal low dose estrogen in the treatment of Overactive Bladder Syndrome at 12 weeks post-treatment initiation. The hypothesis is that low dose intra-vaginal estrogen confers greater benefit than tolterodine in the treatment of Overactive Bladder symptoms. Secondary outcomes were to assess if the addition of the other therapy to the treatment regimen conferred benefit at 24 weeks and 52 weeks.

DETAILED DESCRIPTION:
Lower urinary tract bladder storage symptoms include urinary frequency, urinary urgency, nocturia and urge incontinence. Overactive Bladder (OAB)Syndrome is a condition in which urgency is the predominant symptom with or without urge incontinence and is usually accompanied by frequency and nocturia. The mainstay of treatment of women with OAB syndrome is treatment with anticholinergic medication as well as behavioral therapy. This method of treatment has demonstrated a 60% response rate as reported in the Cochrane Database of Systemic Reviews.

In addition to anticholinergic therapy, vaginal atrophy is often corrected as part of a pharmacologic treatment plan. Vaginal atrophy is a condition this is vastly prevalent in post-menopausal women. It is thought to affect up to 48% of post-menopausal women. Many women with this condition experience vaginal dryness, irritation, painful intercourse, as well as urinary symptoms including dysuria, urgency, frequency, nocturia, incontinence and recurrent urinary tract infections.

Comparison: Tolterodine LA compared to low dose intra-vaginal estrogen cream for the treatment of OAB symptoms

ELIGIBILITY:
Inclusion Criteria:

* Irritative voiding symptoms to include sensory urgency, frequency, urge incontinence, nocturia
* Postmenopausal women with a prior oophorectomy or 1 year from last menstrual period
* Women age 40-90
* Women with hysterectomy with preserved ovaries must be age 55 or greater or have a documented follicle-stimulating hormone (FSH)>40 to ensure post-menopausal status
* Community dwelling
* Ambulatory
* Ability to participate in a 12 month study

Exclusion Criteria:

* Post-void residual volume>150ml
* Glaucoma without ophthalmologist clearance
* Hormone replacement therapy in the past 6 months
* Current anticholinergic treatment
* Breast cancer
* Impaired mental status
* Undiagnosed vaginal bleeding in the past 12 months
* Endometrial thickness on pelvic ultrasound >5mm
* History of thromboembolic event
* Gynecologic cancer
* Untreated urinary tract infection (would be eligible after treatment)
* Stage III pelvic organ prolapse or greater
* Recent diuretic medication changes (one month from change)
* Neurologic condition affecting bladder function (Multiple Sclerosis, Parkinsons, spinal cord injury, spina bifida)
* Congestive heart failure
* Prior pelvic irradiation
* Interstitial cystitis

Ages: 40 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2007-04; Primary Completion 2010-07 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Gerten, M.D., Principal Investigator — Park Nicollette, St. Louis, Minnesota; Holly E. Richter, Ph.D., M.D., Principal Investigator — University of Alabama at Birmingham

REFERENCES:
- [Derived] Ellington DR, Szychowski JM, Malek JM, Gerten KA, Burgio KL, Richter HE. Combined Tolterodine and Vaginal Estradiol Cream for Overactive Bladder Symptoms After Randomized Single-Therapy Treatment. Female Pelvic Med Reconstr Surg. 2016 Jul-Aug;22(4):254-60. doi: 10.1097/SPV.0000000000000256. PMID 26945271

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Extended Release Tolterodine: 4 mg Tolterodine po daily for 12 weeks
  At 12 Weeks, the subjects were offered the addition of the alternative therapy with follow-up at 24 and 52 weeks.
- Group 2: Intra Vaginal Estradiol Cream: 0.5 grams of Intra vaginal estradiol cream nightly for 6 weeks, then twice weekly for 6 weeks.
  At 12 Weeks, the subjects were offered the addition of the alternative therapy with follow-up at 24 and 52 weeks
Period: Treatment For 12 Weeks
Arm/Group | Group 1: Extended Release Tolterodine | Group 2: Intra Vaginal Estradiol Cream
Started | 30 | 28
Completed | 25 | 25
Not Completed | 5 | 3
Not completed — Lost to Follow-up | 4 | 1
Not completed — Family Issues | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Treatment From 12 Weeks To 24 Weeks
Arm/Group | Group 1: Extended Release Tolterodine | Group 2: Intra Vaginal Estradiol Cream
Started | 14 (We included data only from participants that had complete data sets.) | 14 (We included data only from participants that had complete data sets.)
Completed | 14 | 14
Not Completed | 0 | 0
Period: Treatment From 24 Weeks to 52 Weeks
Arm/Group | Group 1: Extended Release Tolterodine | Group 2: Intra Vaginal Estradiol Cream
Started | 11 (We included data only from participants that had complete data sets.) | 14
Completed | 11 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Extended Release Tolterodine: 4 mg Tolterodine po daily for 12 weeks
- Group 2: Intra Vaginal Estradiol Cream: 0.5 grams of Intra vaginal estradiol cream nightly for 6 weeks, then twice weekly for 6 weeks
- Total: Total of all reporting groups
Arm/Group | Group 1: Extended Release Tolterodine | Group 2: Intra Vaginal Estradiol Cream | Total
Number analyzed (Participants) | 30 | 28 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (6) | 60 (2) | 61.5 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 28 | 58
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Evaluate Subjective Patient Change in Irritative Urinary Symptoms as Measured by the Overactive Bladder Questionnaire (OAB-q) Symptom Bother Score
Description: The first part of the OAB-q consists of eight questions assessing symptom bother with a possible score from 0 to 100 with a higher score indicating greater symptom bother.
Time Frame: From baseline through 12 Weeks of Intervention
Population: A baseline measure was achieved for Group 1 with 30 patients and Group 2 with 28 patients. At the 12 week measurement period, we were unable to analyze 5 patients in Group 1 (leaving 25 patients) and unable to analyze 3 patients in Group 2 (leaving 25 patients). These participants left for reasons identified in the Participant Flow.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Group 2: Intravaginal Estradiol Cream: 0.5 grams of Intravaginal estradiol cream nightly for 6 weeks, then twice weekly for 6 weeks
Arm/Group | Group 1: Extended Release Tolterodine | Group 2: Intravaginal Estradiol Cream
Number analyzed (Participants) | 30 | 28
units on a scale
  Baseline | 65.4 (15.3) | 61.6 (20.0)
  12 Weeks: number analyzed (Participants) | 25 | 25
  12 Weeks | 46.7 (23.4) | 45.4 (21.0)
Statistical Analysis 1: Comparison: Group 1: Extended Release Tolterodine vs Group 2: Intravaginal Estradiol Cream; Test type: Superiority; p = .45, t-test, 2 sided

2. Secondary Outcome: Evaluate Subjective Patient Change in Irritative Urinary Symptoms as Measured by the Health Related Quality of Life (HRQL)
Description: Assessment made using the Health Related Quality of Life (HRQL) portion of the OAB-q. The second part of the OAB-q, the HRQL consists of 25 questions that assesses HRQL which addresses coping, concern, sleep and social interaction where the scoring scale is from 0 to 100 with a higher score indicating a better quality of life.
Time Frame: From baseline through 12 Weeks of Intervention
Population: In Group 1, we were unable to analyze 5 patients and in Group 2 we were unable to analyze 3 patients. These participants left for reasons identified in the Participant Flow.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Extended Release Tolterodine: Tolterodine LA: Tolterodine LA 4 mg once daily for 52 weeks
- Intravaginal Estradiol Cream: Estrace Intravaginal Cream: 17-B estradiol cream 0.5 grams nightly for 6 weeks then two times weekly for 46 weeks
Arm/Group | Extended Release Tolterodine | Intravaginal Estradiol Cream
Number analyzed (Participants) | 30 | 28
units on a scale
  Baseline | 53.1 (22.2) | 60.9 (22.5)
  12 weeks: number analyzed (Participants) | 25 | 25
  12 weeks | 66.0 (26.6) | 69.8 (18.2)

3. Secondary Outcome: Evaluate Subjective Patient Change in Irritative Urinary Symptoms
Description: Assessment measured using the Patient Global Impression of Improvement (PGI-I), patient perception of improvement. The PGI-I is a transition scale that is a single question asking the patient to rate their urinary tract condition now, as compared with how it was prior to before beginning treatment on a scale from 1 being very much better to 7 being very much worse.
  Frequencies of each response was reported. Each level achieved (movement towards 1), is considered an improvement.
Time Frame: From baseline through 12 Weeks of Intervention
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Group 1: Extended Release Tolterodine | Group 2: Intravaginal Estradiol Cream
Number analyzed (Participants) | 25 | 25
participants
  Very Much Better | 3 | 0
  Much Better | 8 | 7
  A Little Better | 8 | 12
  No Change | 5 | 5
  A Litlle Worse | 1 | 0

4. Secondary Outcome: Subjective Patient Change in Irritative Urinary Symptoms
Description: This was measured using the Patient Satisfaction Questionnaire (PSQ). The PSQ consists of a single question, "How satisfied are you with your progress since your treatment" in which the 3 possible responses are "completely satisfied," "somewhat satisfied," and "not satisfied." The goal of treatment was to move all participants to "completely satisfied.
Time Frame: From baseline through 12 Weeks of Intervention
Population: In Group 1, we were unable to analyze 5 patients and in Group 2 we were unable to analyze 3 patients. For this outcome ONLY, 1 patient from each Group were not available to obtain the measurements from this questionnaire. Therefore the overall number of participants analyzed for this outcome is less than other outcomes. Please see Participant Flow.
Measure: Number; unit: participants
Groups:
- Extended Release Tolterodine LA: An anti-muscarinic drug that is used for symptomatic treatment of urinary incontinence.
  Extended Release Tolterodine LA: Tolterodine LA 4 mg once daily for 52 weeks
- Intravaginal Estradiol Cream: For topical application to the vaginal area to treat symptoms of urgency or irritation with urination.
  Intravaginal Estradiol Cream: 17-B estradiol cream 0.5 grams nightly for 6 weeks then two times weekly for 46 weeks
Arm/Group | Extended Release Tolterodine LA | Intravaginal Estradiol Cream
Number analyzed (Participants) | 24 | 24
participants
  Completely Satisfied | 5 | 3
  Somewhat Satisfied | 13 | 13
  Not Satisfied | 6 | 8

5. Secondary Outcome: Subjective Patient Change in Irritative Urinary Symptoms As Measured By the 3-Day Voiding Diary
Description: Number of voids and accidents/leakage per 3 day diary. A void is a voluntary and intentional event. An accident is involuntary and unintentional.
Time Frame: From baseline through 12 weeks of Intervention
Population: 25 patients in each group completed voiding diary at baseline. 21 patients completed the voiding diary at 12 weeks in the Tolterodine group (complete diary). 25 patients in the estradiol group completed diary at 12 weeks. Incomplete diaries were not included in our analysis.
Measure: Mean (Standard Deviation); unit: events
Groups:
- Group 2: Intravaginal Estradiol Cream: 0.5 grams of Intravaginal estradiol cream nightly for 6 weeks, then twice weekly for 6 weeks.
  At 12 Weeks, the subjects were offered the addition of the alternative therapy with follow-up at 24 and 52 weeks
Arm/Group | Group 1: Extended Release Tolterodine | Group 2: Intravaginal Estradiol Cream
Number analyzed (Participants) | 21 | 25
events
  Number of voids | 30.4 (11.6) | 26.4 (10.5)
  Number of voids 12 week follow-up | 26.3 (9.7) | 24.6 (10.2)
  Number of accidents/leakage | 10.8 (11.4) | 11.9 (10.5)
  Number of accidents/leakage at 12 weeks | 7.2 (10.6) | 7.7 (8.1)

6. Secondary Outcome: Subjective Patient Change in Irritative Urinary Symptoms
Description: as for outcome 1
Time Frame: Baseline to 24 weeks
Population: At 24 weeks, only 14 patients from Group 1 & 2 had complete data sets. Those without complete data sets were not included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Group 1: Extended Release Tolterodine + Intravaginal Estradiol: After 12 weeks of therapy, participants were offered the alternative therapy in addition to their current therapy. They continued with the 4 mg Tolterodine po daily for 12 weeks and added the 0.5 grams intravaginal estradiol twice per week for 24 weeks.
- Group 2: Intravaginal Estradiol Cream + Tolterodine: 0.5 grams of Intravaginal estradiol cream nightly for 6 weeks, then twice weekly for 6 weeks + 4 mg Tolterodine daily
  (At 12 Weeks, the subjects were offered the addition of the alternative therapy with follow-up at 24 and 52 weeks.)
Arm/Group | Group 1: Extended Release Tolterodine + Intravaginal Estradiol | Group 2: Intravaginal Estradiol Cream + Tolterodine
Number analyzed (Participants) | 14 | 14
units on a scale | -25.4 (11.6) | -28.7 (20.5)

7. Secondary Outcome: Subjective Patient Change in Irritative Urinary Symptoms
Description: as for outcome 2
Time Frame: Baseline to 24 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Group 1: Extended Release Tolterodine + Intravaginal Estradiol: After 12 weeks of therapy, participants were offered the alternative therapy in addition to their current therapy . They continued with the 4 mg Tolterodine po daily for 12 weeks and added the 0.5 grams intravaginal estradiol twice per week for 24 weeks.
Arm/Group | Group 1: Extended Release Tolterodine + Intravaginal Estradiol | Group 2: Intravaginal Estradiol Cream + Tolterodine
Number analyzed (Participants) | 14 | 14
units on a scale | 19.3 (16.8) | 20.9 (15.8)

8. Secondary Outcome: Subjective Patient Change in Irritative Urinary Symptoms as Indicated by the Patient Global Impression of Improvement (PGI-I)
Description: Assessment measured using the Patient Global Impression of Improvement (PGI-I), patient perception of improvement. The PGI-I is a transition scale that is a single question asking the patient to rate their urinary tract condition now, as compared with how it was prior to before beginning treatment on a scale from 1 being very much better to 7 being very much worse. Each level achieved(movement towards 1), is considered an improvement.
Time Frame: Baseline through 24 weeks
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Groups:
- Group 2: Intravaginal Estradiol Cream + Tolterodine: 0.5 grams of Intravaginal estradiol cream nightly for 6 weeks, then twice weekly for 6 weeks + 4 mg Tolterodine daily
  (After 12 weeks of therapy, participants were offered the alternative therapy in addition to their current therapy.)
Arm/Group | Group 1: Extended Release Tolterodine + Intravaginal Estradiol | Group 2: Intravaginal Estradiol Cream + Tolterodine
Number analyzed (Participants) | 14 | 14
percentage of participants | 77 | 77

9. Secondary Outcome: Subjective Patient Change in Irritative Urinary Symptoms as Indicated by the Patient Satisfaction Questionnaire (PSQ)
Description: As measured by the Patient Satisfaction Questionnaire (PSQ). The PSQ consists of a single question, "How satisfied are you with your progress since your treatment" in which the 3 possible responses are "completely satisfied," "somewhat satisfied," and "not satisfied." The goal of treatment was to move all participants to "completely satisfied.
Time Frame: Baseline through 24 weeks
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Groups:
- Group 2: Intravaginal Estradiol Cream + Tolterodine: 0.5 grams of Intravaginal estradiol cream nightly for 6 weeks, then twice weekly for 6 weeks+ 4 mg Tolterodine daily
  (After 12 weeks of therapy, participants were offered the alternative therapy in addition to their current therapy.)
Arm/Group | Group 1: Extended Release Tolterodine + Intravaginal Estradiol | Group 2: Intravaginal Estradiol Cream + Tolterodine
Number analyzed (Participants) | 14 | 14
percentage of participants | 88 | 88

10. Secondary Outcome: Subjective Patient Change in Irritative Urinary Symptoms
Description: as for outcome 1
Time Frame: Baseline through 52 weeks
Population: At 52 weeks, only 11 patients in Group 1 and 14 patients from Group 2 had complete data sets. Those without complete data sets were not included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Group 1: Extended Release Tolterodine + Intravaginal Estradiol: After 12 weeks of therapy, participants were offered the alternative therapy in addition to their current therapy. They continued with the 4 mg Tolterodine po daily for 12 weeks and added the 0.5 grams intravaginal estradiol twice per week for 52 weeks
- Intravaginal Estradiol Cream + Tolterodine: Intravaginal estradiol Cream: 17-B estradiol cream 0.5 grams nightly for 6 weeks then two times weekly for 46 weeks+ 4 mg Tolterodine daily
  At 12 Weeks, the subjects were offered the addition of the alternative therapy with follow-up at 24 and 52 weeks.
Arm/Group | Group 1: Extended Release Tolterodine + Intravaginal Estradiol | Intravaginal Estradiol Cream + Tolterodine
Number analyzed (Participants) | 11 | 14
units on a scale | -23.4 (15.6) | -31.3 (24.3)

11. Secondary Outcome: Subjective Patient Change in Irritative Urinary Symptoms
Description: as for outcome 2
Time Frame: Baseline through 52 weeks
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1: Extended Release Tolterodine + Intravaginal Estradiol | Group 2: Intravaginal Estradiol Cream
Number analyzed (Participants) | 11 | 14
units on a scale | 26.8 (20.5) | 19.7 (25.1)

12. Secondary Outcome: Subjective Patient Change in Irritative Symptoms as Indicated by the Patient Global Impression of Improvement (PGI-I)
Description: as for outcome 8
Time Frame: Baseline through 52 weeks
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Groups:
- Group 2: Intravaginal Estradiol Cream: 0.5 grams of Intra vaginal estradiol cream nightly for 6 weeks, then twice weekly for 6 weeks.
  At 12 Weeks, the subjects were offered the addition of the alternative therapy with follow-up at 24 and 52 weeks
Arm/Group | Group 1: Extended Release Tolterodine + Intravaginal Estradiol | Group 2: Intravaginal Estradiol Cream
Number analyzed (Participants) | 11 | 14
percentage of participants | 85 | 85

13. Secondary Outcome: Subjective Patient Change in Irritative Urinary Symptoms as Indicated by the Patient Satisfaction Questionnaire (PSQ)
Description: As measured by the Patient Satisfaction Questionnaire (PSQ).The PSQ consists of a single question, "How satisfied are you with your progress since your treatment" in which the 3 possible responses are "completely satisfied," "somewhat satisfied," and "not satisfied." The goal of treatment was to move all participants to "completely satisfied.
Time Frame: Baseline through 52 Weeks
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: Extended Release Tolterodine + Intravaginal Estradiol | Group 2: Intravaginal Estradiol Cream
Number analyzed (Participants) | 11 | 14
percentage of participants | 84 | 84

ADVERSE EVENTS:
Time Frame: From Baseline through 52 weeks of Intervention
Groups:
- Group 1: Extended Release Tolterodine: 4 mg Tolterodine po daily for 12-weeks
  At 12 Weeks, the subjects were offered the addition of the alternative therapy with follow-up at 24 and 52 weeks.
- Group 2: Intra Vaginal Estradiol Cream: 0.5 grams of Intra vaginal estradiol cream nightly for 6 weeks, then twice weekly for 6 weeks
  At 12 Weeks, the subjects were offered the addition of the alternative therapy with follow-up at 24 and 52 weeks.
Arm/Group | Group 1: Extended Release Tolterodine | Group 2: Intra Vaginal Estradiol Cream
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/28
Other Adverse Events (participants affected / at risk) | 17/30 | 6/28
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Extended Release Tolterodine (N=30) | Group 2: Intra Vaginal Estradiol Cream (N=28)
xerostomia (General disorders) | 17 (17) | 6 (6) — Xerostomia (also termed dry mouth as a symptom or dry mouth syndrome) is dryness in the mouth (xero- + stom- + -ia), which may be associated with a change in the composition of saliva, or reduced salivary flow, or have no identifiable cause.
Constipation (Gastrointestinal disorders) | 10 (10) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-30): https://cdn.clinicaltrials.gov/large-docs/94/NCT00465894/Prot_SAP_000.pdf